CLINICAL TRIAL: NCT01893697
Title: The Influence of Posture on Airway Diameter, Resistance and Airflow Distribution in Healthy Subjects
Status: Completed | Type: Observational
Sponsor: University Hospital, Antwerp (Other)
Responsible Party: Principal Investigator, Wilfried De Backer, Prof. Dr. W De Backer, University Hospital, Antwerp
Other Study IDs: RESPT_2013_01
Record Dates: First submitted 2013-06-27; First posted 2013-07-09 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: Healthy Participants

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Healthy Participants: HRCT scan in a specific postural position
  Interventions: Other: HRCT scan in a specific postural position

INTERVENTIONS:
Other: HRCT scan in a specific postural position — HRCT Scan taken in supine and lateral position

SUMMARY:
FRI could give the opportunity to investigate the possible effect of a lateral posture on airway diameter and airflow distributions. This physiological study in healthy subjects may help to identify the role of positioning as an aid in airway clearance techniques for patients with respiratory diseases.

DETAILED DESCRIPTION:
Many respiratory diseases require a physiotherapeutic treatment that focusses on clearance of excessive mucus from the airways.

The underlying physiological hypothesis why those mucus clearance techniques are effective is based on the development of an optimal expiratory airflow velocity that applies shearing forces on the mucus at the inner surface of the airway. These shearing forces eventually lead to displacement of mucus to the central airways were it could be evacuated.To accomplish optimal velocity with the same expiratory airflow, it is necessary to decrease the airway diameter and hence increase in the airflow velocity. In other words, the airway diameter and resistance are important factors to take into account in mucus clearance techniques.

In many mucus clearance techniques, postural position is used to facilitate this clearance. Clinical trials in patients with chronic obstructive pulmonary disease (COPD) and cystic fibrosis where they combined clearance techniques with different postural positions showed to be effective.

The influence of posture has been evaluated in the lateral decubitus position and resulted in a greater clearance of mucus in the depended lung. The authors suggested that this may be due to a better deflation of the depended lung that is favored by 3 forces: gravity, mediastinum weight and pressure of abdominal viscera on the infra lateral lung. Deflation of this lung leads not only to a decrease in lung volume, but also results in a decrease in airway diameter. Nevertheless, it is not known to what extend this decrease in diameter occurs in a lateral position. Furthermore, an optimal expiratory flow must be retained in the underlying lung at lower lung volumes. These regional changes in the underlying lung cannot be measured by for example classic lung function tests since these test are not sensitive enough. Indeed, Washko et. al. found no significant changes of overall residual volume (RV), total lung capacity (TLC) and vital capacity (VC) between the different positions in healthy subject.

However, Functional respiratory imaging (FRI) is able to assess the regional changes in healthy subjects. This 3D imaging technique in combination with computational fluid dynamics (CFD) is accurate in calculating regional changes such as airway diameter, volume and resistance. In addition, repetitive FRI measures are able to assess lobar expansion, which is an indirect measure of airflow distribution in a specific part of the lung.

ELIGIBILITY:
Inclusion Criteria:

1. Men or female patients age > 18
2. No respiratory disease in the days prior to the enrollment
3. Able to perform a lung function tests
4. Motivated to participate.
5. Written informed consent from the subject prior to the participation

Exclusion Criteria:

1. Serious co-morbidity which would interfere with the examinations
2. One or multiple CT scans of the chest during the last year.
3. Deformities or complications preventing patients to maintain side lying position during the scanning procedure

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy subjects
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2013-04; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Functional Respiratory Imaging | 1 study visit (1 day)
  A low dose 3D spiral high resolution computed tomography (HRCT) scan will be taken on 2 volumes TLC and functional residual capacity (FRC) in both supine and lateral decubitus position. Image post processing is performed to look at local changes in airway or lobar volume [liter] and airway resistance [kiloPascal.seconds/liter] distribution in the lung

CONTACTS AND LOCATIONS:
Overall Officials: Wilfried De Backer, MD PhD, Principal Investigator — University Hospital, Antwerp
Locations (1):
- UZA, Antwerp, Edegem, Belgium

REFERENCES:
- [Derived] Ides KM, De Backer WA, Lanclus M, Leemans G, Dierckx W, Lauwers E, Vissers D, Steckel J, De Backer JW. The effect of posture on airflow distribution, airway geometry and air velocity in healthy subjects. BMC Pulm Med. 2022 Dec 15;22(1):477. doi: 10.1186/s12890-022-02276-5. PMID 36522658